CLINICAL TRIAL: NCT07101328
Title: BAF_FRontier-1, A First-in-Human, Phase 1 Trial to Assess Safety, Tolerability, and Preliminary Efficacy of LY4152199, a B-cell Activation Factor Receptor (BAFF-R) T-Cell Engager Bispecific Antibody in Adult Participants With Previously Treated B-cell Malignancies
Brief Title: A Study of LY4152199 in Participants With Previously Treated B-cell Cancers (BAF_FRontier-1 )
Acronym: BAF_FRontier-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27701; J6N-MC-JUCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma, Non-Hodgkin; B-cell Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular
Keywords: Bispecific antibody; Non-Hodgkin Lymphoma; B-cell activating factor; B- cell activating factor receptor (BAFFR); BAFFR
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Dose Escalation (Cohort A DLBCL and FL) (Experimental): Escalating doses of LY4152199 administered intravenously (IV)
  Interventions: Drug: LY4152199 - IV
- Phase 1: Dose Optimization (Cohort B1 DLBCL) (Experimental): Two or more doses of LY4152199 (evaluated during dose escalation) administered IV
  Interventions: Drug: LY4152199 - IV
- Phase 1: Dose Optimization (Cohort B2 FL) (Experimental): Two or more doses of LY4152199 (evaluated during dose escalation) administered IV
  Interventions: Drug: LY4152199 - IV

INTERVENTIONS:
Drug: LY4152199 - IV — Administered by IV infusion

SUMMARY:
The purpose of this study is to find the best dose of the drug and measure the safety and efficacy of LY4152199 in participants with previously treated B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Estimated life expectancy of greater than or equal to (≥)12 weeks as judged by the Investigator.
* Participants with select tumor types must have measurable or assessable disease as defined below:
* Must have at least 1 bi-dimensionally measurable lesion or in the absence of measurable lymphadenopathy, documentation of bone marrow involvement.
* Must be able to comply with inpatient/outpatient treatment, laboratory monitoring, and required clinic visits for the duration of trial participation.
* Must have adequate organ function.
* Must have failed or were intolerant to at least 2 prior lines of therapy appropriate for available treatment for the specific B-cell malignancy

Exclusion Criteria:

All Participants

* Known or suspected central nervous system (CNS) involvement by systemic lymphoma.
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Any unresolved toxicities from prior therapy greater than National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade 2 at the time of starting trial treatment except for alopecia.
* Autologous stem cell transplantation within 100 days of this study for post autologous transplant individuals.
* Residual symptoms of neurotoxicity or cytopenias from prior chimeric antigen receptor T-cell therapy (CAR-T) or bispecifics. Exception: Cytopenia related to prior CAR-T or bispecifics allowed if they meet the adequate organ function criteria.
* Known or suspected history of macrophage activation syndrome or hemophagocytic lymphohistiocytosis (HLH).
* Active second malignancies, unless in remission, with life expectancy greater than 2 years with Sponsor approval.
* History of autoimmune disease
* Significant cardiovascular disease
* Active uncontrolled systemic bacterial, viral, fungal, or parasitic infection (except for fungal nail infection), or other clinically significant active disease process
* Vaccination with a live vaccine within 4 weeks prior to signing informed consent form (ICF).
* Have current or had a history of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins).
* Prior treatment with B-cell activating factor receptor (BAFF-R) directed therapies (e.g., monoclonal antibody, CAR-T or bispecific antibody). This exclusion criterion does not apply to participants seeking retreatment.
* Pregnant and/or planning to breastfeed during the trial or within 90 days of the last dose of study intervention.
* Known hypersensitivity to any component or excipient of LY4152199.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - Number of Participants with Dose Limiting Toxicities (DLT) of LY4152199 | Approximately 35 days

SECONDARY OUTCOMES:
Phase 1 - Pharmacokinetics (PK): Area under the Concentration versus Time Curve (AUC) of LY4152199 | Baseline up to approximately 91 weeks
Phase 1- PK: Maximum drug Concentration (Cmax) of LY4152199 | Baseline up to approximately 91 weeks
Phase 1 - Overall Response Rate (ORR): Percentage of Participants with Best Overall Response of Complete Response (CR) or Partial Response (PR) | Baseline up to approximately 4 years until disease progression or start of new anti-cancer therapy
  Assessed by the Investigator per disease-specific response criteria as appropriate or death due to any cause, whichever occurs first
Phase 1 - Duration of Response (DOR) | Baseline up to approximately 4 years until disease progression or start of new anti-cancer therapy
  Time between the date of first documented response (CR or PR) to the date of first disease progression or death due to any cause, whichever occurs first
Phase 1- Time to Response (TTR) | Baseline up to approximately 4 years until disease progression or start of new anti-cancer therapy
  Time from first dose date (or randomization date for the dose optimization cohort) to the date of first documented response (CR or PR)
Phase 1 - Progression Free Survival (PFS) | Baseline up to approximately 4 years until disease progression or start of new anti-cancer therapy
  Time from first dose date (or randomization date for the dose optimization cohort) to the date of first documented disease progression or death due to any cause, whichever occurs first
Phase 1- Disease Control Rate (DCR) | Baseline up to approximately 4 years until disease progression or start of new anti-cancer therapy
  Percentage of efficacy-evaluable participants who achieved a BOR of CR, PR, or stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (50):
- United States (23):
  - City of Hope, Duarte, California
  - University of Colorado Denver - School of Medicine - Anschutz Medical Campus, Aurora, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New York University (NYU) Clinical Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Swedish Cancer Institute (SCI), Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - The Alfred Hospital, Melbourne, VIC
  - Linear Clinical Research, Nedlands
- Canada (3):
  - Lady Davis Institute for Medical Research Jewish General Hospital, Montreal
  - University Health Network (UHN) - Princess Margaret Cancer Centre, Toronto
  - BC Cancer - Vancouve, Vancouver
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Center for Cancer and Organ Diseases - Rigshospitalet, Copenhagen
- France (2):
  - CHU de Lille - Hopital Claude Huriez, Lille
  - AP-HP Hopital Saint-Louis, Paris
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - LMU Klinikum Muenchen-Campus Grosshadern, München
  - Universitaetsklinikum Muenster, Münster
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant Orsola, Bologna
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Istituto Clinico Humanitas, Rozzano
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - Okayama University Hospital, Okayama
  - Cancer Institute Hospital of JFCR, Tokyo
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - AIDPORT Sp. z o.o., Skorzewo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No